CLINICAL TRIAL: NCT03533413
Title: A Modified Technique of Combined Fluoroscopy and CT Guided Thermal Radiofrequency Ablation of Thoracic Dorsal Root Ganglia in Intractable Pain Associated With Thoracic Malignancies: A Randomized Clinical Trial
Brief Title: Combined Fluoroscopy and CT Guided Radiofrequency Ablation of Thoracic Dorsal Root Ganglia in Severe Thoracic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, lecturer of anesthesia ,critical care and pain medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Raafat-Ehab.combined
Record Dates: First submitted 2018-04-22; First posted 2018-05-23 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Cancer-related Problem/Condition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional:Combined CT-fluroscopy (Active Comparator): Combined CT-fluroscopic radiofrequency ablation of thoracic dorsal root ganglia.
  Interventions: Procedure: combined CT-fluroscopy
- Interventional: standard fluroscopy (Active Comparator): Fluroscopic radiofrequency ablation of thoracic dorsal root ganglia.
  Interventions: Procedure: standard fluroscopy

INTERVENTIONS:
Procedure: combined CT-fluroscopy — Radiofrequency ablation of thoracic dorsal root ganglia guided by combined CT-Fluroscopy
  Arms: Interventional:Combined CT-fluroscopy
Procedure: standard fluroscopy — Radiofrequency ablation of thoracic dorsal root ganglia guided by standard fluroscopy only
  Arms: Interventional: standard fluroscopy

SUMMARY:
In the current study, extra-guidance other than conventional fluoroscopy - will be integrated to improve the success of the transforaminal approach to the thoracic dorsal root ganglia (DRG). The investigators hypothesize that joining CT scan with fluoroscopy to guide RF ablation through the transforaminal route may enhance its efficacy and safety in relieving the intractable pain associated with chest malignancies. The current study aimed to compare the results of thermal radiofrequency ablation (TRFA) of the thoracic DRG under combined CT and fluoroscopy guidance with the classic standard fluoroscopy technique.

DETAILED DESCRIPTION:
Thoracic pain represents about 3-5% of pain clinics' visitors worldwide .Post-thoracotomy pain occurs in 30%-50% of patients undergoing thoracotomy .Interventional therapies include epidural or intrathecal drug injection, intercostal nerve block, sympathectomy, rhizotomy, and percutaneous cervical cordotomy. Rhizotomy refers to the selective segmental destruction of the dorsal sensory rootlets to interrupt pain perception by the spinal cord. This could be accomplished either neurosurgically, chemically or using selective percutaneous procedures such as cryoanalgesia and radiofrequency (RF) ablation.There are many technical difficulties in approaching the deep-seated thoracic dorsal root ganglia (DRG) through the transforaminal route.The spine is kyphotic - with the tip at T6 - and slightly scoliotic to the right side even in normal subjects . Spinous processes are acute, especially at T5-T8 level. Besides, broad and wide laminae together with narrow intervertebral foramina are other obstacles .The intervertebral foramina are further masked by the facet joints and the crowdedness of the costovertebral and the costotransverse joints .For all these factors, more guidance - other than conventional fluoroscopy - may improve the success of the transforaminal approach to the thoracic DRG. The investigators hypothesize that joining CT scan with fluoroscopy to guide RF ablation through the transforaminal route can enhance its efficacy and safety in relieving the intractable pain of chest malignancies. The current study aimed to compare the results of thermal radiofrequency ablation (TRFA) of the thoracic DRG under combined CT and fluoroscopy guidance with the classic standard fluoroscopy technique.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or more
* suffering from chronic moderate-to-severe pain ( VAS score ≥ 40 mm)
* due to malignancy involving the chest and pain was refractory to the maximally tolerated dose of opioids for at least four weeks. Malignancies included : lung cancer, pleural mesothelioma, chest wall tumors and metastatic deposits of the chest.

Exclusion Criteria:

* sepsis, coagulopathy
* malignant epidural invasion
* distorted local anatomy
* severe cardiorespiratory compromise
* neuropsychiatric illness
* history of drug dependence and known allergy to contrast media or the used medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
pain relief. | 12 weeks follow up
  Pain intensity measured by visual analog scale (VAS).It measures the pain intensity and percentage of pain relief.The investigators used 100 mm horizontal scale with left zero end representing no pain and right 100 end representing worst pain.Scores ranging 0-39 reflect mild pain , 40-69 moderate pain and 70-100 severe pain.

SECONDARY OUTCOMES:
patient satisfaction. | 12 weeks
  The secondary outcome measure will be assessed using patient satisfaction with the patient global impression of changes (PGIC).It measures the degree of patient overall satisfaction after the performed procedure. It includes 7 domains ranging from 1 to 7. the first domain indicates that the patient is very much improved while the 7th domain indicates that he is very much worsened by the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
It will be a shared team work study during which all the investigators will have equally distributed roles.

REFERENCES:
- [Derived] Reyad RM, Ghobrial HZ, Shaker EH, Reyad EM, Shaaban MH, Hashem RH, Darwish WM. Modified technique for thermal radiofrequency ablation of Thoracic dorsal root ganglia under combined fluoroscopy and CT guidance: a randomized clinical trial. BMC Anesthesiol. 2019 Dec 18;19(1):234. doi: 10.1186/s12871-019-0906-4. PMID 31852438
- See also: clinical journal of pain — https://www.ncbi.nlm.nih.gov/pubmed/8788580